CLINICAL TRIAL: NCT06907043
Title: A Phase 1/2, Open-label, Multicenter, Dose-escalation, and Dose-Optimization Study to Evaluate the Safety, Tolerability, and Activity of EIK1004 (IMP1707) as Monotherapy in Participants With Advanced Solid Tumors
Brief Title: A Study of PARP1 Selective Inhibitor, EIK1004 (IMP1707) in Participants With Advanced Solid Tumors.
Acronym: EIK1004-001
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eikon Therapeutics (Industry)
Collaborators: Impact Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EIK1004-001(IMP1707-101); IMP1707-101 (Other: IMPACT Therapeutics Inc.)
Record Dates: First submitted 2025-03-22; First posted 2025-04-02 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Advanced Solid Tumors
Keywords: EIK1004; IMP1707; Advanced/recurrent/metastatic pancreatic adenocarcinoma; Brain metastases; Advanced HER2-negative breast adenocarcinoma; Recurrent HER2-negative breast adenocarcinoma; metastatic HER2-negative breast adenocarcinoma
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Intervention Model Description: Groups of participants are assigned to receive interventions for dose escalation in up to 7 cohorts.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Part 1 (Experimental): EIK1004 (IMP1707) monotherapy; oral tablet(s) daily (except for the single-dose period). Participants will receive escalating doses of EIK1004 (IMP1707) until progressive disease or discontinuation.
  Interventions: Drug: EIK1004-001 (IMP1707-001)

INTERVENTIONS:
Drug: EIK1004-001 (IMP1707-001) — PARP1 selective inhibitor

SUMMARY:
This study will evaluate the safety, tolerability, and preliminary efficacy of EIK1004 (IMP1707) in participants with recurrent advanced/metastatic breast cancer, ovarian cancer, metastatic castrate resistant prostate cancer (mCRPC) and pancreatic cancer with deleterious/suspected deleterious mutations of select homologous recombination repair (HRR) genes.

Condition or disease Intervention/treatment Phase Advanced Solid Tumors Drug: EIK1004 (IMP1707) Phase 1/Phase 2

DETAILED DESCRIPTION:
This study will evaluate the safety, tolerability and preliminary efficacy of EIK1004 (IMP1707) as monotherapy in patients with recurrent, advanced/metastatic solid tumors. The study consists of 2 parts: Dose escalation and dose optimization.

In dose escalation (Part1), the study will identify the maximum tolerated dose (MTD) or maximum achievable dose (MAD) in solid tumor.

In dose optimization (Part 2), the study will further evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and anti-tumor activity of select doses of EIK1004 (IMP1707)

ELIGIBILITY:
• Breast cancer: must have received at least one prior chemotherapy in neoadjuvant/adjuvant/metastatic setting, must have received hormonal therapy if HR+, HGSOC or high grade endometrioid EOC, fallopian tube or primary peritoneal cancer; must have received at least one prior platinum-based chemotherapy for advanced disease.

mCRPC with ongoing ADT, must have received NHA and up to 1 prior line of taxane chemotherapy; Pancreatic cancer, must have prior 1L therapy

* Age ≥ 18 years at the time of informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status ≤1
* Adequate organ function
* Life expectancy ≥ 12 weeks
* Should have evaluable disease as defined by RECIST1.1 and/or CA125 or PSA
* Female subjects of childbearing potential and male subjects must agree to use an effective method of contraception from study entry up to 6 months after the last dose of EIK1004 (IMP1707)
* Deleterious or suspected deleterious germline or somatic mutations of select HRR genes
* Up to 1 prior line of PARP inhibitor containing treatment

CNS Inclusion Criteria:

* Untreated CNS metastases (measurable and/or non-measurable) not needing immediate local therapy.
* Previously treated CNS metastases

Key Exclusion Criteria:

* Any investigational or approved anti-cancer therapies administered within 28 days/ before the first dose of EIK1004 (IMP1707)
* Have received prior PARP1 selective inhibitors
* Mean resting QTcF > 470 ms or QTcF < 340 ms
* Infections

  - An active hepatitis B/C infection
* Any known predisposition to bleeding
* Unable to swallow oral medications OR have malabsorption syndrome or any other uncontrolled gastrointestinal condition that might impair the bioavailability

CNS Exclusion Criteria

* Any untreated brain lesions > 2.0 cm in size.
* Ongoing use of systemic corticosteroids for control of symptoms of CNS metastases < 7 days prior to the first dose of study treatment or requirement for > 10 mg prednisone/day.
* Any brain lesion requiring immediate local therapy, including (but not limited to) a lesion in an anatomic site where an increase in size or possible treatment-related edema may pose risk to the participant (eg, brain stem lesions).
* Known, symptomatic leptomeningeal disease.
* Have poorly controlled seizures.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants who experience a Dose-Limiting Toxicity (DLT) | (Timeframe: up to 28 days)
  A DLT is defined as an event with toxicity including the type, severity, time of onset, time of resolution, and the probable association with study treatment that are not due to pre-existing conditions as defined by the Common Terminology Criteria for Adverse Events Version 5.0 (CTCAE 5.0). The number of participants who experience a DLT will be reported.
Number of participants with adverse events, treatment emergent adverse events or serious adverse events | (Time Frame: 1 month post last dose of EIK1004 (IMP1707)
  Number of participants reporting adverse events or serious adverse events which include any abnormal clinical events, laboratory assessments outside of normal clinical range, abnormal vital signs observed, and any abnormal ECG parameters

SECONDARY OUTCOMES:
Pharmacokinetic parameters of EIK1004 (IMP1707) | Through study completion, up to 3 years
  Peak plasma concentration (Cmax)
Pharmacokinetic parameters of EIK1004 (IMP1707) | Time Frame: Through study completion, up to 3 years
  Area under the curve (AUC) will be defined
Objective Response (OR) | Through study completion, up to 3 years
  Defined as participants who have a complete response [CR] or Participants who have a partial response [PR] by RECIST 1.1 (Solid tumor) and RANO-BM (brain metastasis), or CA-125 response per GCIG criteria (ovarian cancer), or PSA response per PCWG3 criteria.

OTHER OUTCOMES:
Pharmacodynamic changes due to EIK1004 (IMP1707) | Through study completion, up to 3 years
  Cytokines will be measured using an ELISA assay. The concentration of cytokines in plasma samples collected from patients is being measured and will be reported as a quantified value (e.g ng/mL).
  The fold change in plasma cytokines over baseline will be measured and the relative change compared to pre-dose/baseline numbers.

CONTACTS AND LOCATIONS:
Overall Officials: Yawei Zhang, MD, Study Director — Eikon Therapeutics
Locations (10):
- United States (6):
  - Sarah Cannon Research Institute at HealthOne, Denver, Colorado
  - Florida Cancer Center, Lake Mary, Florida
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - MD Anderson, Houston, Texas
  - NEXT Oncology, San Antonio, Texas
  - NEXT Virginia, Fairfax, Virginia
- PASO Medical, Frankston, Victoria, Australia
- China (3):
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Cancer Hospital of Shandong First Medical University(Shandong Cancer Institute, Shandong Cancer Hospital), Jinan, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai